CLINICAL TRIAL: NCT06638814
Title: HEmorrhoidAl Disease in Inflammatory Bowel Disease: a Multicenter Prospective Cohort Study
Acronym: HEAD-IBD-II
Status: Not yet recruiting | Type: Observational
Sponsor: Treviso Regional Hospital (Network)
Responsible Party: Principal Investigator, Ugo Grossi, MD PhD, Assistant Professor of Surgery, Treviso Regional Hospital
Other Study IDs: HEAD-IBD-II
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: IBD (Inflammatory Bowel Disease); Hemorrhoid; Safety; Sugery; Surgery Related Complications Rate
Keywords: HEAD-IBD-II; Hemorrhoidal disease; IBD; Surgery
MeSH Terms: conditions — Inflammatory Bowel Diseases; Hemorrhoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients who will undergo surgery for hemorrhoidal disease after the diagnosis of IBD: All patients with an established diagnosis of IBD who will undergo surgery for HD from January to December 2025 and followed-up for at least 1 year post-operatively will be prospectively included. Data on patient demographics and clinical characteristics, operative details and clinical outcomes will be collected.

SUMMARY:
Patients who will undergo surgery for HD after the diagnosis of IBD over a 12-month period will be enrolled across Europe.

Primary objective of this study is to determine the safety and effectiveness of surgical treatments for HD in a large multicenter cohort of IBD patients.

Secondary aim is to identify factors that may affect clinical and surgical outcomes.

DETAILED DESCRIPTION:
To date, there is no consensus in the scientific literature regarding the exact indications for surgery for hemorrhoidal disease (HD) in patients with inflammatory bowel disease (IBD). The HEAD-IBD-II study is a multicenter, prospective cohort designed to evaluate the safety and effectiveness of surgical treatments for hemorrhoidal disease (HD) in patients with inflammatory bowel disease (IBD). This study aims to collect contemporary, real-world data from multiple hospitals across various countries, focusing on the surgical management of HD in this unique patient population. The study will include adult patients with a confirmed diagnosis of Crohn's disease or ulcerative colitis who undergo surgery for HD.

The data collection process will involve detailed records of patient demographics, pre-operative status, operative techniques, and post-operative outcomes, with a specific focus on short-, medium-, and long-term surgical and clinical results. The study will track outcomes such as postoperative complications, recurrence of symptoms, IBD flare-ups, and anal continence.

In addition, factors such as surgical volume, techniques employed, and individual patient characteristics will be analyzed to identify variables that may impact the outcomes. The study is designed to generate hypotheses and explore variability in current practices, thereby highlighting areas in need of further investigation through randomized controlled trials.

All patient data will be collected anonymously through a secure electronic case report form (eCRF), and results will be disseminated according to the STROBE guidelines for observational studies. Ethical approval will be obtained from participating institutions, and all patients will provide informed consent prior to inclusion. The study is expected to improve the understanding of surgical approaches to HD in IBD patients and potentially guide future clinical recommendations.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 years and above;
* established diagnosis of Crohn's disease or ulcerative colitis at the time of surgery for hemorrhoidal disease;
* planned surgery for hemorrhoidal disease during the study period, including hemorrhoidectomy (open, close or submucosal), transanal hemorrhoidal dearterialization, hemorrhoidal laser procedure, stapled hemorrhoidopexy).

Exclusion Criteria:

* previous surgery for hemorrhoidal disease other than office-based treatments (e.g., sclerotherapy injection, rubber band ligation);
* active perianal disease at the time of surgical intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo surgery for hemorrhoidal disease after the diagnosis of IBD will be enrolled in several centers across the European territory.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety and effectiveness of surgical treatments for hemorrhoidal disease | 12 months from surgery
  Data on patient demographics and clinical characteristics, operative details, and clinical and surgical outcomes will be collected.
  The surgical outcomes will include: length of hospital stay, 30-day readmission, and post-operative complications at medium- (6 months) and long-term (12 months) follow-up.
  The clinical outcomes will include: IBD flare, defined according to standard scores (i.e., partial Mayo score for ulcerative colitis and Harvey-Bradshaw Index for Crohn's disease) and need for therapeutic change or dose escalation during the 6 months after surgery, new onset of perianal disease, anal continence status at last follow-up.

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared due to concerns related to patient confidentiality and the sensitive nature of the clinical data involved in this study. Although the data will be anonymized, the sharing of IPD may still pose risks regarding patient privacy. Furthermore, the study's results will be shared in aggregate form through peer-reviewed publications, ensuring transparency and dissemination of the findings without compromising individual data privacy.

REFERENCES:
- [Background] Grossi U, Gallo G, Di Tanna GL, Bracale U, Ballo M, Galasso E, Kazemi Nava A, Zucchella M, Cinetto F, Rattazzi M, Felice C, Zanus G. Surgical Management of Hemorrhoidal Disease in Inflammatory Bowel Disease: A Systematic Review with Proportional Meta-Analysis. J Clin Med. 2022 Jan 28;11(3):709. doi: 10.3390/jcm11030709. PMID 35160159